CLINICAL TRIAL: NCT05619276
Title: Acute Intervention to Assess the Impact of Practical Strategies to Facilitate a Balanced and Healthy Diet
Brief Title: Acute Intervention to Assess the Impact of Practical Strategies for Healthy Eating
Acronym: PORTIONS-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: University of Bristol (Other); University of Roma La Sapienza (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PC171-172; 2022.121 (Other: University of Navarra Research Ethics Committee)
Record Dates: First submitted 2022-10-24; First posted 2022-11-16 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2023-11

CONDITIONS: Overweight and Obesity; Healthy Diet
Keywords: Portion control tools; Food portion size
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: The study involves two stages. During stage 1 (control condition) all participants will use conventional kitchen utensils to self-serve and condiment a laboratory meal. During stage 2 (experimental condition) all participants will use an experimental set of tools to self-serve and condiment the same meal as in stage 1. The two stages will always follow the same order, control first and then experimental. The before and after design was chosen as the study aims to explore the acute effect of the implementation of portion control utensils in the same individual, avoiding carry-over effects due to learning from using the experimental tool.
Who Masked: Participant
Masking Description: The study will be advertised as research on practical strategies to facilitate a balanced and healthy diet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard serving utensil toolkit (Active Comparator): Participants will self-serve and condiment a cold meal in the laboratory using standard kitchen utensils, including 2 nylon serving spoons and a simple glass oil dispenser. Participants will complete an eye-tracking test before eating, and will fill in questionnaires and provide blood samples during and after the meal. At 2h post-meal, they will complete a computerized memory reconstruction task related to the meal. After leaving the laboratory participants will keep a food diary, and will complete an on-line learning test before bedtime.
  Interventions: Device: Standard serving utensil toolkit
- Optimised portion-control toolkit (Experimental): Participants will self-serve and condiment a cold meal in the laboratory using an optimised portion control toolkit. This toolkit will include two calibrated serving spoons, one for vegetables (slotted) and one for starch (solid), and a calibrated oil dispenser. Both spoons have a volume capacity of 155 ml with a 121 ml mark. The oil dispenser has a volume capacity of 250ml and allows pre-portioning of the oil via a sucking device in amounts ranging from 5-20 millilitres, 1-3 teaspoons or 0.5 to 1 tablespoon, prior to serving. Participants will complete an eye-tracking test before eating, and will fill in questionnaires and provide blood samples during and after the meal. At 2h post-meal, they will complete a computerized memory reconstruction task related to the meal. After leaving the laboratory participants will keep a food diary, and will complete an on-line learning test before bedtime.
  Interventions: Device: Optimsed portion-control toolkit

INTERVENTIONS:
Device: Standard serving utensil toolkit — Serving a meal using standard kitchen utensils (100% of subjects experiment with these tools first)
  Other Names: Standard serving spoon set and standard oil dispenser
  Arms: Standard serving utensil toolkit
Device: Optimsed portion-control toolkit — Serving a meal using optimised, portion-control utensils (100% of subjects experiment with these tools second)
  Other Names: Calibrated serving spoon set and calibrated oil dispenser
  Arms: Optimised portion-control toolkit

SUMMARY:
Obesity has reached epidemic proportions globally, alongside its associated comorbidities including cardiovascular diseases, diabetes and cancer. Effective weight management strategies are thus paramount to improve the population´s health. One of the key causes of obesity lies in excessive energy consumption derived from eating too large portions of food. In this context, practical tools to control portion size represent a promising, cost-effective strategy.

This study will investigate whether using an optimized portion-control toolkit to consume a meal under controlled laboratory conditions has a positive effect on the nutritional quality of the meal as well as any benefits in physiological, cognitive, affective and behavioural outcomes.

The study will involve 40 volunteers with overweight or obesity who will attend two lunch sessions at the Center for Nutrition Research of the University of Navarra (Spain) on two different days. At each session, participants will be invited to self-serve and eat a lunch from a cold buffet. On day one, participants will self-serve and season their food using control tools (conventional kitchen serving spoons and oil dispenser). On day two, participants will self-serve the same foods as on day one but using experimental tools (calibrated portion-control serving spoons and calibrated oil dispenser). A set of cognitive tests will be completed before, during and after the meal.

Conventional and experimental tools will be compared in terms of the following variables: meal portion size and energy density, cognitive effort while serving food, cephalic and intestinal satiety responses, appetite sensations, energy adjustment post-meal, awareness of the quantities of the previously consumed foods and recalibration of portion size norms. Additionally, the study will explore acceptance for and intention to use the optimized portion control toolkit, as well as intention to change eating habits.

It is expected that the findings from this study will shed light into the cognitive and physiological processes associated with portion control. It may also help to explain individual variations in the responses to obesogenic environments, which will hopefully lead to improved personalized interventions.

DETAILED DESCRIPTION:
Study justification:

The prevalence of obesity and associated health-risks (e.g. cardiovascular disease, diabetes and cancer) continues to increase across the globe, raising the need for effective weight management strategies to improve the population´s health. High rates of obesity respond at least in part, to the current obesogenic environment that prompts people to overeat both in terms of energy and amount. In this context, access to practical tools that can help individuals control their portion sizes represent a promising, cost-effective strategy. However, urging people to "eat less" of all foods might be challenging as individuals are used to consume a certain volume of food to feel satisfied. Instead, a more effective approach may be to help people lower the energy density of their meals through the increase in the amount of fruits and vegetables in their diet at the expense of high energy density foods, such as foods rich in fat and starch. Portion-control plates and serving utensils, designed to measure the appropriate amounts and proportions of main food groups (e.g. starch, protein and vegetables), can actually facilitate this shift. Our recent systematic review (https://pubmed.ncbi.nlm.nih.gov/34207492/) found that portion-control plates in particular were the most promising tools to regulate intake and develop healthier eating habits. However, some of the studies conducted up to date have explored the effect of different portion control tools in combination with other weight management strategies, making it difficult to determine the impact of these instruments on their own. The design of the tools may also negatively affect success if instruments don´t fit the user´s lifestyle and eating routines. Individual characteristics such as sex and BMI have also been found to modulate the success of portion control tools. Therefore, optimizing the current tools is needed to achieve a wider impact.

Specific aims:

The primary goal of the present study is to investigate the acute effects of using a portion control tableware toolkit, optimized based on our previous quantitative and qualitative work with portion control tableware, in people with overweight and obesity. The intervention will be conducted under controlled laboratory conditions in order to obtain proof of concept of the toolkit efficacy before application into field studies. The secondary goal is to gain knowledge on the cognitive and physiological mechanisms involved in portion size regulation mediated by portion control tools.

It is expected that the findings from this study will shed light into the cognitive and physiological processes associated with portion control. It may also help to explain individual variations in the responses to obesogenic environments, which will hopefully lead to improved personalized interventions. The ultimate goal is to develop effective, easy, attractive and affordable strategies that could help individuals prevent overeating.

Study design:

This will be a non-randomized within-subjects laboratory study which will involve two sessions, of approximately 3 - hour duration each, conducted at lunchtime at the Center for Nutrition Research of the University of Navarra (Pamplona) on two different days, with a 7 to 11 day wash-out period. At each session, participants will be invited to self-serve and eat a lunch from a cold buffet in the laboratory. On day one, participants will self-serve and season their food using control tools (conventional kitchen serving spoons and oil dispenser). On day two, participants will be invited to self-serve the same foods as on day one but using experimental tools (calibrated portion control serving spoons and calibrated oil dispenser). On both days, the food will be served on a standard (25 cm in diameter), white dish without markings or illustrations, and participants will eat using standard cutlery. A set of cognitive tests will be completed before, during and after the meal. All participants will receive a give-away tool in compensation for their time.

Study procedures:

* 100 mm visual analogue scales (VAS) will be used for hunger-satiety assessment prior to the meal intake, immediately after finishing the meal and at 30, 60, 90 and 120 minutes after finishing the meal.
* Blood extractions will be carried out at 0 (fasting), and then 7, 12, 32, 62 and 92 minutes after commencing the lunch. Blood levels of glucose, insulin, pancreatic polypeptide and total ghrelin will be used as biomarkers of satiety/hunger.
* A wearable Tobii eye-tracking device will be used during the self-serving activity to infer cognitive effort associated to the serving task from total and average fixation durations, fixation count, time to first fixation and pupil dilation.
* A computerized memory reconstruction task will be completed by participants 120 minutes after beginning meal intake to measure the accuracy of the participants' recall of the food amounts consumed. Specifically, visual representation through selected images of the previously consumed amounts (recalled portion size) will be compared to actual amounts consumed after the use of each set of tools (consumed portion sizes).
* A food diary will be kept by participants up to bed-time after they leave the laboratory on each study day to monitor energy and macronutrient intake, plus compensatory eating behaviour.
* A computerized learning reconstruction task, aimed at recreating a balanced meal using images of foods, will be completed by participants before going to bed.
* Questionnaires will be used to evaluate the intention to change one's eating habits after using the experimental tools, perceived cognitive effort when using experimental tools, toolkit acceptance, and to compare participants' habitual portion sizes (portion size norms) with the ones selected in the laboratory.
* An observation task will be conducted at the end of visit 2, to collect participants' opinions about 3 additional portion-control utensils developped/chosen based on our previous qualitative study (a multi-compartment lunchbox, a portion-control melanine dish and a measuring cup for dry food).

Experimental buffet:

The experimental buffet has been designed to include foods from each of the main food groups in line with the USDA MyPlate model. The foods include: vegetables (cherry tomatoes, green leaves and bell pepper), protein (cooked chopped chicken breasts, canned tuna and mozzarella cheese pearls) a starchy food (cooked quinoa and pasta). Chickpeas are also included as starchy food although they contain some protein. Fruit including apples, oranges and canned pineapple, is included as optional dessert. Complimentary bread, condiments (olive oil, salt, and pepper) and non-carbonated water will also be offered.

All foods and water will be served cold (or at room temperature) on separate trays set up in a buffet-style and in sufficient amounts to allow eating until comfortably full and to avoid ceiling effects (e.g. at least double the amount of the average portion). To standardize the two study conditions, participants will be asked to select the same foods on both laboratory visits. Each participant will choose his/her own experimental meal during the screening session, thereby preventing any unnecessary food waste.

Recruitment and Screening:

The sample size for this study was estimated using the open source software GPower. For a 2-sided paired comparison, a sample of 34 completers would allow detection of significant between-conditions differences, with alpha 0.05 and 80% power, in variables related to selected portion size (main outcome measure: consumed carbohydrate portion size), cognitive effort, and cephalic and intestinal satiety responses. Assuming a 15% drop-out (based on an observed 10% rate in our previous study) the recruitment target will be 40 healthy adults with overweight or obesity. Whenever possible, a balanced representation of men and women will be ensured, so that neither sex constitutes more than 60% (or less than 40%) of the sample. Potential participants will be recruited through advertisements in the local press, through social media, university newsletters, at health and community centres, pharmacies, shops, schools, etc., and from the volunteer database from the Center for Nutrition Research of the University of Navarra.

Initial verification of the inclusion/exclusion criteria will be performed via a telephone interview. If the initial criteria are met, candidates will be sent via email a link and ID code to complete the Eating Attitudes Test (EAT-26) and the Perceived Stress Scale (PSS-14) online, via Google Forms. Those who meet the EAT-26 and PSS-14 criteria (see Eligiblity Criteria section) will be invited to the screening session in the laboratory for anthropometric measurements, experimental food tasting, and an eye-tracking familiarization test.

Assessment:

The following questionnaires will be administered to collect data for later sample description and analysis of potential variables that could influence eating habits and hence study results:

* Socio-demographic questionnaire.
* NEO Five-Factor Inventory (NEO-FFI), to assess the central domains of normal personality
* Profile of mood states (POMS), to explore potential impact of emotions on eating behavior.
* Trait meta-mood scale (TMMS-24), to measure of emotional intelligence
* Three-factor eating questionnaire (TFEQ), to measure the three dimensions of human eating behavior (dietary restraint, disinhibition and hunger)
* Beverage consumption habits (BPS), to explore beverage portion size awareness and consumption habits.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 65 years
* BMI between 27.5 and 39 kg/m-sq, except for Asian participants (BMI 26 to 39 kg/m-sq)
* Good gastrointestinal health
* Good visual acuity or wearing contact lenses
* Regular eating habits (i.e. consuming lunch and dinner at least 5 days a week)
* Liking of at least one of the foods from the three major categories (vegetables, protein, and starch)
* Willingness to provide blood samples
* Availability to attend two clinical visits at lunch time

Exclusion Criteria:

* Malnutrition (including dehydration; anaemia; blood donation within less than 3 months)
* Gastrointestinal disorders
* Eating disorders (a score of 20 or more in the EAT-26)
* Elevated stress levels (a score of 27 or more in the PSS-14)
* Need to wear glasses to self-serve food
* Being on a diet to gain or lose weight (leading to >7.5% body weight change in the last 3 months)
* Food allergies or restrictions impacting food choices at the buffet meal (including veganism)
* Active medical conditions like diabetes, cancer, epilepsy, memory loss impacting on food behaviour and/or body weight
* Taking medications affecting appetite, body weight, memory or sight, except if the person has been on a stable dose for the past 3 months and no symptoms have been experienced
* Using a pacemaker/other electronic medical device that may interfere with the eye tracking equipment or software
* Smokers, drinkers, athletes and pregnant or lactating women
* Knowledge that can affect the results of the study (e.g., nutritionists/dietitians, those with previous training in eating behaviour research)
* Participation in the preceeding qualitative study.

Menstrual cycle in women will not be controlled for but day of last menstruation in pre-menopausal women will be recorded. Post-menopausal women will not be excluded; however, this detail will be noted at screening, with an individual's menopausal status (pre, peri or post).

Candidates working shifts may be eligible if they are able to attend a clinical visit at least 12 hours since the last shift, to ensure they have sufficient sleep and their appetite sensations are not altered.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline (standard tookit condition) in consumed portion size of carbohydrate under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Grams of consumed carbohydrate

SECONDARY OUTCOMES:
Change from baseline (standard tookit condition) in consumed portion size of protein under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Grams of consumed protein
Change from baseline (standard tookit condition) in consumed portion size of vegetables under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Grams of consumed vegetables
Change from baseline (standard tookit condition) in consumed portion size of fat under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Grams of consumed fat
Change from baseline (standard tookit condition) in consumed portion size of fibre under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Grams of consumed fibre
Change from baseline (standard tookit condition) in served portion size of carbohydrate under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Grams of served carbohydrate
Change from baseline (standard tookit condition) in served portion size of protein under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Grams of served protein
Change from baseline (standard tookit condition) in served portion size of vegetables under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Grams of served vegetables
Change from baseline (standard tookit condition) in served portion size of fat under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Grams of served fat
Change from baseline (standard tookit condition) in served portion size of fibre under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Grams of served fibre
Change from baseline (standard tookit condition) in post-prandial blood glucose at 7 min under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Blood glucose levels at 7 min post-meal
Change from baseline (standard tookit condition) in post-prandial blood glucose at 12 min under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Blood glucose levels at 12 min post-meal
Change from baseline (standard tookit condition) in post-prandial blood glucose at 32 min under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Blood glucose levels at 32 min post-meal
Change from baseline (standard tookit condition) in post-prandial blood glucose at 62 min under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Blood glucose levels at 62 min post-meal
Change from baseline (standard tookit condition) in post-prandial blood glucose at 92 min under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Blood glucose levels at 92 min post-meal
Change from baseline (standard tookit condition) in post-prandial blood insulin at 7 min under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Blood insulin levels at 7 min post-meal
Change from baseline (standard tookit condition) in post-prandial blood insulin at 12 min under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Blood insulin levels at 12 min post-meal
Change from baseline (standard tookit condition) in post-prandial blood insulin at 32 min under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Blood insulin levels at 32 min post-meal
Change from baseline (standard tookit condition) in post-prandial blood insulin at 62 min under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Blood insulin levels at 62 min post-meal
Change from baseline (standard tookit condition) in post-prandial blood insulin at 92 min under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Blood insulin levels at 92 min post-meal
Change from baseline (standard tookit condition) in post-prandial blood pancreatic polypeptide at 7 min under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Blood pancreatic polypeptide levels at 7 min post-meal
Change from baseline (standard tookit condition) in post-prandial blood pancreatic polypeptide at 12 min under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Blood pancreatic polypeptide levels at 12 min post-meal
Change from baseline (standard tookit condition) in post-prandial blood pancreatic polypeptide at 32 min under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Blood pancreatic polypeptide levels at 32 min post-meal
Change from baseline (standard tookit condition) in post-prandial blood pancreatic polypeptide at 62 min under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Blood pancreatic polypeptide levels at 62 min post-meal
Change from baseline (standard tookit condition) in post-prandial blood pancreatic polypeptide at 92 min under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Blood pancreatic polypeptide levels at 92 min post-meal
Change from baseline (standard tookit condition) in post-prandial blood ghrelin at 7 min under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Blood total ghrelin levels at 7 min post-meal
Change from baseline (standard tookit condition) in post-prandial blood ghrelin at 12 min under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Blood total ghrelin levels at 12 min post-meal
Change from baseline (standard tookit condition) in post-prandial blood ghrelin at 32 min under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Blood total ghrelin levels at 32 min post-meal
Change from baseline (standard tookit condition) in post-prandial blood ghrelin at 62 min under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Blood total ghrelin levels at 62 min post-meal
Change from baseline (standard tookit condition) in post-prandial blood ghrelin at 92 min under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Blood total ghrelin levels at 92 min post-meal
Total serving time (min) | Clinical Investigation Day 1
  Duration of the serving time for the meal (min) at the first serving
Total serving time (min) | Clinical Investigation Day 2
  Duration of the serving time for the meal (min) at the first serving
Visual fixation time (sec) | Clinical Investigation Day 1
  Duration of the visual fixation time while serving the meal (sec) at the first serving
Visual fixation time (sec) | Clinical Investigation Day 2
  Duration of the visual fixation time while serving the meal (sec) at the first serving
Pupil dilation (mm) | Clinical Investigation Day 1
  Dilation of the pupil while serving the meal (mm) at the first serving
Pupil dilation (mm) | Clinical Investigation Day 2
  Dilation of the pupil while serving the meal (mm) at the first serving

OTHER OUTCOMES:
Change from baseline (standard tookit condition) in fasting blood glucose under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Fasting blood glucose levels
Change from baseline (standard tookit condition) in fasting blood insulin under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Fasting blood insulin levels
Change from baseline (standard tookit condition) in fasting blood pancreatic polypeptide under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Fasting blood pancreatic polypeptide levels
Change from baseline (standard tookit condition) in fasting blood ghrelin under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Fasting blood ghrelin levels
Portion tool Acceptance | Clinical Investigation Day 1
  Average 5-Pt Likert scores for portion tool acceptance, ease of use, perceived effectiveness and intention to use (previously piloted questionnaire), after self-serving of the meal and before meal consumption. An average score of 1 or 2 indicates low acceptance, 3 neutral, and 4 or 5 high acceptance.
Portion tool Acceptance | Clinical Investigation Day 2
  Average 5-Pt Likert scores for portion tool acceptance, ease of use, perceived effectiveness and intention to use (previously piloted questionnaire), after self-serving of the meal and before meal consumption. An average score of 1 or 2 indicates low acceptance, 3 neutral, and 4 or 5 high acceptance.
Change from baseline (standard toolkit condition) in Subjective cognitive effort, under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Subjective cognitive effort (self-constructed questionnaire), after self-serving of the meal and before meal consumption. A higher score indicates a greater perceived effort in conducting the task.
Change from baseline (standard toolkit condition) in Intention to change habits (Priming), under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Intention to change eating habits and to maintain the newly acquired habits (self-constructed questionnaire), after self-serving of the meal and before meal consumption. A higher score indicates a stronger intention to change and/or perceived capacity to achieve the desired change.
Area Under the Curve for subjective hunger | Clinical Investigation Day 1
  Area Under the Curve for hunger levels calculated from the 100 mm visual analogue scale scores for hunger before the meal and at 30, 60, 90 and 120 min after meal initiation (validated questionnaire)
Area Under the Curve (AUC) for subjective hunger | Clinical Investigation Day 2
  AUC for hunger levels calculated from the 100 mm visual analogue scale scores for hunger before the meal and at 30, 60, 90 and 120 min after meal initiation (validated questionnaire)
Area Under the Curve for subjective fullness | Clinical Investigation Day 1
  Area Under the Curve for fullness levels calculated from the 100 mm visual analogue scale scores for fullness before the meal and at 30, 60, 90 and 120 min after meal initiation (validated questionnaire)
Area Under the Curve for subjective fullness | Clinical Investigation Day 2
  Area Under the Curve for fullness levels calculated from the 100 mm visual analogue scale scores for fullness before the meal and at 30, 60, 90 and 120 min after meal initiation (validated questionnaire)
Area Under the Curve for subjective thirst | Clinical Investigation Day 1
  Area Under the Curve for thirst levels calculated from the 100 mm visual analogue scale scores for thirst before the meal and at 30, 60, 90 and 120 min after meal initiation (validated questionnaire)
Area Under the Curve for subjective thirst | Clinical Investigation Day 2
  Area Under the Curve for thirst levels calculated from the 100 mm visual analogue scale scores for thirst before the meal and at 30, 60, 90 and 120 min after meal initiation (validated questionnaire)
Area Under the Curve for subjective prospective intake | Clinical Investigation Day 1
  Area Under the Curve for prospective intake levels calculated from the 100 mm visual analogue scale scores for thirst before the meal and at 30, 60, 90 and 120 min after meal initiation (validated questionnaire)
Area Under the Curve for subjective prospective intake | Clinical Investigation Day 2
  Area Under the Curve for prospective intake levels calculated from the 100 mm visual analogue scale scores for thirst before the meal and at 30, 60, 90 and 120 min after meal initiation (validated questionnaire)
Area Under the Curve for nausea | Clinical Investigation Day 1
  Area Under the Curve for nausea levels calculated from the 100 mm visual analogue scale scores for thirst before the meal and at 30, 60, 90 and 120 min after meal initiation (validated questionnaire)
Area Under the Curve for nausea | Clinical Investigation Day 2
  Area Under the Curve for nausea levels calculated from the 100 mm visual analogue scale scores for thirst before the meal and at 30, 60, 90 and 120 min after meal initiation (validated questionnaire)
Expected satiety for the meal | Clinical Investigation Day 1
  100 mm visual analogue scale scores for expected satiety of the meal (published scale), after self-serving of the meal, before meal consumption. A higher score indicates that the meal is perceived as more satiating.
Expected satiety for the meal | Clinical Investigation Day 2
  100 mm visual analogue scale scores for expected satiety of the meal (published scale), after self-serving of the meal, before meal consumption. A higher score indicates that the meal is perceived as more satiating.
Portion size norms for meal components | Clinical Investigation Day 1
  100 mm VAS scores for how much the served portion of the whole meal, starch, vegetables and protein differs from an habitual portion (published questionnaire), at 30 min after meal initiation. A score above 50 mm indicates that the participant's habitual portion size is larger than the portion size being evaluated.
Portion size norms for meal components | Clinical Investigation Day 2
  100 mm visual analogue scale scores for how much the served portion of the whole meal, starch, vegetables and protein differs from an habitual portion (published questionnaire), at 30 min after meal initiation. A score above 50 mm indicates that the participant's habitual portion size is larger than the portion size being evaluated.
Liking | Clinical Investigation Day 1
  100 mm visual analogue scale scores for liking of the meal (pre-piloted scale), at 30 min after meal initiation. A higher score indicates higher liking for the meal.
Liking | Clinical Investigation Day 2
  100 mm visual analogue scale scores for liking of the meal (pre-piloted scale), at 30 min after meal initiation. A higher score indicates higher liking for the meal.
Change from baseline (standard toolkit condition) in post-lunch energy intake, under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Energy (kcal) intake during the the 8 h following the laboratory visit, calculated from food data registered in an estimated food diary (published method)
Change from baseline (standard toolkit condition) in post-lunch energy compensation, under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Percent energy compensation during the the 8 h following the laboratory visit, calculated from food data registered in an estimated food diary (published method)
Change from baseline (standard toolkit condition) in memory reconstruction error, under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Percent error between actual (g) and recalled (g) portion sizes for the foods consumed at the laboratory lunch, using a computerised task at 120 min after meal initiation (published method)
Change from baseline (standard toolkit condition) in portion size learning, under the portion-control toolkit condition | Clinical Investigation Day 1, Clinical Investigation Day 2
  Percent error between recreated portion sizes (g) and recommended portion sizes (g) for a sample of representative foods, using an on-line computerised task, before bed time (unpublished method)
Socio-demographic profile | Screening visit
  Descriptive profile composed of self-reported age, gender, educational level, ethnic origin, marital status, household composition, employment, meal composition and patterns, main shopper
Body weight | Screening visit
  Weight (kg) measured wearing indoor clothing
Height | Screening visit
  Height (cm) measured without shoes
Body Mass Index (BMI) | Screening visit
  Adipositiy index calculated as body weight (kg) divided by squared height (in m)
Personality | Screening visit
  Score in the NEO-Five Factor Inventory 60 item validated questionnaire. The score for each central domain of normal personality defined by the Five-Factor Model of personality (neuroticism, extraversion, conscientiousness, agreeableness, and openness to experience) is calculated. A higher score on a scale assessing a certain personality domain indicates a stronger expression of traits associated with this particular domain.
Emotional intelligence | Screening visit (on-line questionnaire at home)
  Score in the Trait Meta-Mood Scale-24 validated questionnaire. The score for three different dimensions of emotional intelligence are calculated. To obtain a score for each factor, items 1 to 8 are added for the emotional attention factor, items 9 to 16 for the emotional clarity factor, and items 17 to 24 for the emotional repair factor.
Mood profile | Screening visit (on-line questionnaire at home)
  Score in the Profile of Mood States validated questionnaire. The score for six different dimensions of mood (tension, anger, fatigue, depression, confusion, and vigour) is calculated. A higher score on a scale assessing a certain mood dimension indicates a stronger expression of associated feelings. The resulting scores will range from -24 to 177, with lower scores indicative of people with more stable mood profiles.
Test meal liking | Screening visit
  Combined 100 mm visual analogue scale scores for liking of the test meal components
Test meal familiarity | Screening visit
  Combined 100 mm visual analogue scale scores for familiarity with the test meal components
Risk for eating disorders | Pre-screening (on-line questionnaire at home)
  Score in the Eating Attitudes Test-26, ranging from 0-78 points, validated by Garner et al., 1982. Scores above 20 suggest risk for presence of potential eating disorders.
Risk for high stress levels | Pre-screening (on-line questionnaire at home)
  Score in the Perceived Stress Scale validated questionnaire. Scores ranging from 0 to 13 suggest low stress, scores ranging from 14 to 24 suggest moderate stress, and scores above 27 suggest high perceived stress.
Eating habits profile | Screening
  Profile defined by the combined Restraint (0-21 points), Disihnibition (0-16 points) and Susceptibilty to hunger (0-14 points) sub-scales scores of the Three Factor Eating Questionnaire (TFEQ), validated by Stunkard & Messick, 1985. Restraint values above 11, disinhibition values above 8 and susceptibility to hunger values above 4 are considered worse outcomes (i.e. risk for development of obesity and other eating disorders).
Beverage consumption habits | Screening
  Self-reported consumption habits and awareness of beverage portion size (pre-piloted on-line BPS survey)
Novel portion-control tools opinions | Clinical Investigation Day 2
  Opinions from the participant in regards to the perceived acceptability, usefulness and areas of improvement for a set of novel portion-control tools including a lunchbox, measuring cup and commercial portion-control plate (collected via interview)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Almiron-Roig, PhD, Principal Investigator — University of Navarra
Locations (1):
- University of Navarra, Dept. of Food Science and Physiology, Center for Nutrition Research, Pamplona, Navarre, Spain